CLINICAL TRIAL: NCT06050850
Title: A Healthy Weight Intervention for Family Stress During the Early Phases of ALL Treatment: NOURISH-ALL
Brief Title: Healthy Weight Intervention Families During ALL Treatment: NOURISH-ALL
Acronym: NOURISH-ALL
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Children's Mercy Hospital Kansas City (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Carolyn Bates, PhD, Principal Investigator, Assistant Professor, University of Kansas Medical Center
Other Study IDs: STUDY00002516; 1K08CA279877-01A1 (NIH)
Record Dates: First submitted 2023-09-08; First posted 2023-09-22 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: ALL, Childhood; Behavior, Health
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Health Behavior

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aim 1a: Adapting the NOURISH-ALL Intervention for Families of Youth with ALL (Year 1): The purpose of Aim 1a is to adapt the NOURISH-T intervention to meet the specific needs of families during the early phases of ALL treatment. To achieve this goal, the study will initiate a three-step intervention adaptation process that includes (1) initial integration of cognitive behavioral therapy (CBT) and family systems frameworks, (2) formative assessment with families of youth with ALL, and (3) formative assessment with multidisciplinary experts.
- Aim 1b: Iteratively Refining the NOURISH-ALL Intervention (Year 2): The purpose of Aim 1b is to adaptively refine NOURISH-ALL through sequential testing with individual families during the early phases of ALL treatment, with the goal of optimizing feasibility and acceptability from the family perspective. In line with the ORBIT model, the study will utilize an adaptive approach, similar to the commonly known "PDSA cycle," to maximize responsivity to individual patient/family feedback. Participants will receive NOURISH-ALL and provide feedback throughout the intervention (i.e., after each session and upon intervention completion), which will be iteratively analyzed and incorporated to improve intervention delivery for the next family
  Interventions: Behavioral: NOURISH-ALL
- Aim 2: Pilot Single-Arm Trial of NOURISH-ALL Focused on Participant Engagement (Years 3-5): Pilot testing key components of engagement is critical to optimizing design and methodology of fully powered efficacy trials. The purpose of Aim 2 is to pilot a single-arm trial of the finalized NOURISH-ALL intervention in a sample of families of youth in the early phases of ALL treatment to assess recruitment, retention, and dose received. Results will directly inform the design of the fully powered randomized control trial to test intervention efficacy (R01 application to be submitted in Year 4).
  Interventions: Behavioral: NOURISH-ALL

INTERVENTIONS:
Behavioral: NOURISH-ALL — Our NOURISH-ALL intervention will build on this existing NOURISH-T family based behavioral intervention with families of cancer survivors. The intervention, NOURISH-ALL, will adapt these family-based health promotion strategies to the early ALL treatment context.
  Groups: Aim 1b: Iteratively Refining the NOURISH-ALL Intervention (Year 2); Aim 2: Pilot Single-Arm Trial of NOURISH-ALL Focused on Participant Engagement (Years 3-5)

SUMMARY:
The purpose of this study is to conduct a single arm pilot of the NOURISH-ALL (Nourishing Our Understanding of Role modeling to Improve Support and Health in Acute Lymphoblastic Leukemia) intervention focused on three components of participant engagement. This is a single arm intervention study that involves participation in a 6-session family intervention and three time points of multimethod data collection. The primary outcome is participant engagement, measured as recruitment, retention, and intended dose received.

This study will be conducted over 5 years in three phases:

* Aim 1a: Adapting the NOURISH-ALL Intervention for Families of Youth with ALL (Year 1)
* Aim 1b: Iteratively Refining the NOURISH-ALL Intervention (Year 2)
* Aim 2: Pilot Single-Arm Trial of NOURISH-ALL Focused on Participant Engagement (Years 3-5)

DETAILED DESCRIPTION:
The long-term goal of this work is to establish an efficacious family-based health promotion intervention that curbs excessive weight gain among youth with newly diagnosed acute lymphoblastic leukemia (ALL) by integrating support for family coping with stress during the early phases of treatment.

The objectives of the current study are to adapt an existing family-based health promotion intervention, NOURISH-T, to meet the needs of families of youth in the early phases of ALL treatment (NOURISH-ALL) and (2) assess three key components of engagement in preparation for a fully powered efficacy trial.

NOURISH-T is a 6-session family-based health promotion intervention that has demonstrated improved physical activity (PA), dietary intake, and weight among youth who are cancer survivors. Guided by the ORBIT Model of Behavioral Intervention Development, this study will modify NOURISH-T to fit the early ALL treatment context through a multi-stage adaptation and refinement process. Adaptations will incorporate family systems and cognitive behavioral intervention components to support healthy family coping with diagnosis and treatment stress. Additional, patient-centered adaptations will be informed by semi-structured family input around intervention content and delivery.

The central hypothesis is that this rigorous approach to adaptation will yield an intervention that is feasible, acceptable, and engaging for families of youth with ALL. By incorporating tailored strategies for health promotion during the early phases of ALL treatment, the proposed study seeks to shift clinical practice paradigms to prevent weight-related disparities in treatment outcomes.

Hypothesis:

The central hypothesis is that this rigorous approach to adaptation will yield an intervention that is feasible, acceptable, and engaging for families of youth with ALL.

Aims:

AIM 1: To (a) adapt the NOURISH-T intervention to target the early phases of ALL treatment (NOURISH-ALL) and (b) refine this ALL-tailored intervention for optimal feasibility and acceptability from the patient and family perspective. (Years 1-2) Defining the specific needs of families of youth with newly diagnosed ALL is essential to effectively adapting behavior change interventions to the early phases of ALL treatment. Refining interventions for optimal feasibility and acceptability from the family perspective is critical to successful intervention development.

Aim 1a: Intervention Adaptation. The purpose of Aim 1a is to adapt the NOURISH-T intervention to meet the specific needs of families during the early phases of ALL treatment. To achieve this goal, the study will initiate a three-step intervention adaptation process that includes (1) initial integration of cognitive behavioral therapy (CBT) and family systems frameworks, (2) formative assessment with families of youth with ALL, and (3) formative assessment with multidisciplinary experts.

Aim 1b. Refinement to Optimize Feasibility and Acceptability. The purpose of Aim 1b is to adaptively refine NOURISH-ALL through sequential testing with individual families during the early phases of ALL treatment, with the goal of optimizing feasibility and acceptability from the family perspective. In line with the ORBIT model, the study will utilize an adaptive approach, similar to the commonly known "PDSA cycle," to maximize responsivity to individual patient/family feedback. Participants will receive NOURISH-ALL and provide feedback throughout the intervention (i.e., after each session and upon intervention completion), which will be iteratively analyzed and incorporated to improve intervention delivery for the next family.

AIM 2: To conduct an external pilot single-arm trial of NOURISH-ALL focused on three components of engagement. (Years 3-5). Pilot testing key components of engagement is critical to optimizing design and methodology of fully powered efficacy trials. The purpose of Aim 2 is to pilot a single-arm trial of the finalized NOURISH-ALL intervention in a sample of families of youth in the early phases of ALL treatment to assess recruitment, retention, and dose received. Results will directly inform the design of the fully powered randomized control trial to test intervention efficacy (R01 application to be submitted in Year 4).

ELIGIBILITY:
Inclusion Criteria:

* Children ages 2-12 years old and their primary caregiver ages 18-90
* Child diagnosed with acute lymphoblastic leukemia (ALL)
* Child completed induction phase of therapy and not yet in maintenance phase of therapy
* Primary caregiver and child English language proficient
* Primary caregiver able to provide permission for child to participate in research
* Primary caregiver identifies as being involved with child's oncology care
* Primary caregiver lives with child at least 50% of the time
* Primary oncology provider confirms child is eligible to participate

Exclusion Criteria:

* Primary oncology provider identifies safety concerns regarding the child's participation in the study.

Ages: 2 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Families of youth aged 2-12 years who are newly diagnosed with acute lymphoblastic leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Baseline (Week 0)
  Measured by # enrolled / # eligible
Retention Rate | Post-Intervention (Week 6), Follow-Up (Month 6)
  Measured by # completed intervention / # enrolled
Intended dose received | Post-Intervention (Week 6), Follow-Up (Month 6)
  Measured by # sessions attended / # sessions offered

SECONDARY OUTCOMES:
Child Body Mass Index (BMI) | Baseline (Week 0), Post-Intervention (Week 6), Follow-Up (Month 6)
  Measured by child height and weight
Child Physical Activity | Baseline (Week 0), Post-Intervention (Week 6), Follow-Up (Month 6)
  Measured by Actigraph wGT3x+ activity monitor
Child Sleep | Baseline (Week 0), Post-Intervention (Week 6), Follow-Up (Month 6)
  Measured by Actigraph wGT3x+ activity monitor
Child Dietary Intake | Baseline (Week 0), Post-Intervention (Week 6), Follow-Up (Month 6)
  Total calories, % calories from fat, and other nutrition variables will be measured by Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24)
Family Stress Measures | Baseline (Week 0), Post-Intervention (Week 6), Follow-Up (Month 6)
  Measured by Psychosocial Assessment Tool v3.0 (PAT 3.0)
Family Distress | Baseline (Week 0), Post-Intervention (Week 6), Follow-Up (Month 6)
  Measured by Distress Thermometer (DT)
Body Composition - Bioelectrical Impedance Analysis | Baseline (Week 0), Post-Intervention (Week 6), Follow-Up (Month 6)
  Measured by InBody Scale bioelectrical impedance analysis
Body Composition | Baseline (Week 0), Post-Intervention (Week 6), Follow-Up (Month 6)
  Measured by dual energy x-ray absorptiometry (DXA) scan
Subcutaneous fat | Baseline (Week 0), Post-Intervention (Week 6), Follow-Up (Month 6)
  Skinfold thickness measurement

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Bates, PhD, Principal Investigator — University of Kansas Medical Center; Keith August, MD, Principal Investigator — Children's Mercy Kansas City
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Children's Mercy Kansas City, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: Undecided